CLINICAL TRIAL: NCT05791513
Title: The Effectiveness of Using a Clinical Support Tool in Managing Adolescents With Non-Traumatic Knee Pain (The MAP-Knee Trial): a Stepped-wedge Cluster Randomised Trial
Brief Title: The Effectiveness of Using a Clinical Support Tool in Managing Adolescents With Non-Traumatic Knee Pain
Acronym: MAP-Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Michael Skovdal Rathleff, Professor, Aalborg University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: N-20220043
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Knee Pain Chronic

STUDY DESIGN:
Intervention Model Description: Stepped-wedge randomised trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Using the MAP-Knee Tool (Experimental): The treating clinician will use the MAP-Knee Tool together with the adolescent. The tool includes four separate components: 1) a tool for diagnosing the most common types of non-traumatic knee pain (SMILE), 2) credible explanations of the aetiology and pathogenesis specific to the diagnosis based on multiple methods with an iterative design, 3) a presentation of prognostic factors based on an individual participant data meta-analysis(19), and 4) an option grid that presents the users of the tool with pros and cons of commonly used management options based on a systematic literature search of systematic and narrative reviews within non-traumatic adolescent knee pain. An overarching focus of all components was to support shared decision-making and base decisions on all three pillars of evidence-based medicine: patient values, clinical expertise, and relevant research. Therefore, the tool should not provide the users with definitive answers simply based on available evidence.
  Interventions: Other: Using the MAP-Knee Tool
- Not using the MAP-Knee Tool (Active Comparator): The treating clinician will not use the MAP-Knee Tool in the consultation and will conduct the consultation as per usual practice.
  Interventions: Other: Usual practice

INTERVENTIONS:
Other: Using the MAP-Knee Tool — Using the MAP-Knee Tool
  Arms: Using the MAP-Knee Tool
Other: Usual practice — The consultation between clinician and adolescent is conducted as per usual practice.
  Arms: Not using the MAP-Knee Tool

SUMMARY:
The aim of the stepped-wedge cluster randomised trial is to investigate the effectiveness of using a clinical support tool (The MAP-Knee Tool) in managing adolescents aged 10-19 years with non-traumatic knee pain compared to not using the tool. Six participating hospitals will start to use the tool within 4, 6, or 8 months after recruitment start in a randomised order. We will investigate if using the tool is superior in terms of reducing symptoms compared to not using the tool.

DETAILED DESCRIPTION:
The trial will be designed as a stepped-wedge cluster randomised superiority trial to be conducted across 6 hospital departments across Denmark. Any orthopaedic or similar hospital department in Denmark to which adolescents suffering from non-traumatic knee pain may be referred is eligible for participation. Any medical doctor or physiotherapist employed at either of the study sites who regularly see adolescents with non-traumatic knee pain will be eligible to participate in the trial.

Before crossover occurs at the study site, the adolescents will be treated as usual which is at the discretion of the treating clinician. Based on our current research on the usual care pathway, this will be heterogenous and include advice to wait and see, imaging (most often MRI and x-ray), or a rehabilitation plan for the municipality. After crossing over to using the MAP-Knee Tool, the treating clinician will use the MAP-Knee Tool together with the adolescent. The tool was designed to support the entire consultation from diagnosing the condition (patellofemoral pain, Osgood-Schlatter, Sinding-Larsson-Johansson, growth pain, patellar tendinopathy, or iliotibial band syndrome) to deciding on future management. The MAP-Knee Tool includes four separate components: 1) a tool for diagnosing the most common types of non-traumatic knee pain (SMILE), 2) credible explanations of the aetiology and pathogenesis specific to the diagnosis based on multiple methods with an iterative design, 3) a presentation of prognostic factors based on an individual participant data meta-analysis, and 4) an option grid that presents the users of the tool with pros and cons of commonly used management options based on a systematic literature search of systematic and narrative reviews within non-traumatic adolescent knee pain. An overarching focus of all components was to support shared decision-making and base decisions on all three pillars of evidence-based medicine: patient values, clinical expertise, and relevant research. Therefore, the tool should not provide the users with definitive answers simply based on available evidence. After the initial prototype of the tool including all four components had been made, the investigators performed end-user testing using think-aloud sessions with adolescents suffering from non-traumatic knee pain, adolescents with no history of knee pain, and medical doctors.

ELIGIBILITY:
Inclusion Criteria:

* Having been referred to a hospital due to non-traumatic knee pain
* Age between 10 and 19 years

Exclusion Criteria:

* Knee pain with a traumatic origin
* Lack of ability to cooperate

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 110 (Actual)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
KOOS-Child Pain subscale | During baseline and at the 12-week and 52-week follow-ups
  KOOS-Child consists of 39 items divided into five subscales (Pain, Symptoms, Activities of Daily Living, Sport/Recreation, and Quality of Life) that each range from 0 to 100 with 100 being optimum. This questionnaire has been found to have good psychometric properties and is recommended for children and adolescents suffering from knee disorders.

SECONDARY OUTCOMES:
KOOS-Child Symptoms subscale | During baseline and at the 12-week and 52-week follow-ups
  KOOS-Child consists of 39 items divided into five subscales (Pain, Symptoms, Activities of Daily Living, Sport/Recreation, and Quality of Life) that each range from 0 to 100 with 100 being optimum. This questionnaire has been found to have good psychometric properties and is recommended for children and adolescents suffering from knee disorders.
KOOS-Child Activities of daily living subscale | During baseline and at the 12-week and 52-week follow-ups
  KOOS-Child consists of 39 items divided into five subscales (Pain, Symptoms, Activities of Daily Living, Sport/Recreation, and Quality of Life) that each range from 0 to 100 with 100 being optimum. This questionnaire has been found to have good psychometric properties and is recommended for children and adolescents suffering from knee disorders.
KOOS-Child Sport/recreation subscale | During baseline and at the 12-week and 52-week follow-ups
  KOOS-Child consists of 39 items divided into five subscales (Pain, Symptoms, Activities of Daily Living, Sport/Recreation, and Quality of Life) that each range from 0 to 100 with 100 being optimum. This questionnaire has been found to have good psychometric properties and is recommended for children and adolescents suffering from knee disorders.
KOOS-Child Quality of Life subscale | During baseline and at the 12-week and 52-week follow-ups
  KOOS-Child consists of 39 items divided into five subscales (Pain, Symptoms, Activities of Daily Living, Sport/Recreation, and Quality of Life) that each range from 0 to 100 with 100 being optimum. This questionnaire has been found to have good psychometric properties and is recommended for children and adolescents suffering from knee disorders.
EQ-5D-Y | During baseline and at the 12-week and 52-week follow-ups
  Health-related quality of life will be estimated by the EQ-5D-Youth questionnaire which is an adapted version of the EQ-5D used in an adult population, yet, it still consists of the same five subscales which are mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
Global Rating of Change | At the 12-week and 52-week follow-ups
  This will be used to measure the participants' self-reported recovery on a 7-point Likert scale ranging from "much improved" to "much worse". Participants are categorised as improved if they rate themselves as "much improved" or "improved" (category 6-7) and categorised as not improved if they rate themselves from "slightly improved" to "much worse" (category 1-5).
International Physical Activity Questionnaire short version (IPAQ). | During baseline and at the 12-week and 52-week follow-ups
  The IPAQ is the most used questionnaire for measuring physical activity and consists of 9 items that provide information on the time spent performing vigorous and moderate activities, the time spent walking, and time spent sedentary during the past week. The IPAQ gives an estimate of the total weekly physical activity measured in MET-minutes per week and total minutes spent sitting.
Sports participation | During baseline and at the 12-week and 52-week follow-ups
  Change in sports participation will be explored using a questionnaire in which participants are asked about whether they have participated in leisure sports activities, type of sports activities and weekly frequency.

OTHER OUTCOMES:
Anterior Knee Pain Youth (AKP-Youth) | During baseline and at the 12-week and 52-week follow-ups
  We will use our newly developed questionnaire as a secondary measure of condition severity. The AKP-Youth contains 23 items that are divided into four overarching domains of impact: symptoms, limitations in physical activity, limitations in social activities, and emotional impact of pain.

CONTACTS AND LOCATIONS:
Locations (6):
- Denmark (6):
  - Aalborg Universitetshospital, Aalborg
  - Amager-Hvidovre Hospital, Copenhagen
  - Bispebjerg Hospital, Copenhagen
  - Sportsmedicinsk Center, Frederikshavn
  - Næstved Sygehus, Næstved
  - Vejle Sygehus, Vejle

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon reasonable request.